CLINICAL TRIAL: NCT02777827
Title: A Randomised, Double-Blinded, Double-Dummy, Placebo-Controlled, MultiCentre-, Six-Way, Crossover Study to Assess the Pharmacodynamics, Pharmacokinetics, and Safety of Abediterol Single Dose, Given by Dry Powder Inhaler (DPI) or Pressurised Metered-Dose Inhaler (pMDI), in Patients With Asthma on Inhaled Corticosteroids.
Brief Title: A Single Dose PD & PK Study With Two Formulations of Abediterol in Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D6540C00002
Record Dates: First submitted 2016-04-29; First posted 2016-05-19 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: Abediterol; Dry powder inhaler; Pressured metered-dose inhaler; Pharmacokinetic; Pharmacodynamic; Safety
MeSH Terms: conditions — Asthma | interventions — 5-(2-((6-(2,2-difluoro-2-phenylethoxy)hexyl)amino)-1-hydroxyethyl)-8-hydroxyquinolin-2(1H)-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Abediterol dry powder inhaler 0.156 μg (Experimental): Dry powder for inhalation administered via dry powder inhaler 0.156 μg/inhalation; (1 inhalation)
  Interventions: Drug: Abediterol 0.156 μg
- Abediterol dry powder inhaler 2.5 μg (Experimental): Dry powder for inhalation, administered via dry powder, inhaler 2.5 μg/inhalation; (1 inhalation).
  Interventions: Drug: Abediterol 2.5 μg
- Abediterol pressurised metered-dose inhaler 0.05μg (Experimental): Pressurised metered-dose, inhaler 0.025 μg/puff; (2 puffs).
  Interventions: Drug: Abediterol 0.05 μg
- Abediterol pressurised metered-dose inhaler 0.156 μg (Experimental): Pressurised metered-dose, inhaler 0.078 μg/puff; (2 puffs).
  Interventions: Drug: Abediterol 0.156 μg
- Abediterol pressurised metered-dose inhaler 2.5μg (Experimental): Pressurised metered-dose inhaler 1.25 μg/puff; (2 puffs).
  Interventions: Drug: Abediterol 2.5 μg
- Placebo (Placebo Comparator): Pressurised metered-dose inhaler (2 puffs) and Dry powder for inhalation administered via dry powder inhaler (1 inhalation).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Abediterol 0.156 μg — Dry powder for inhalation
  Arms: Abediterol dry powder inhaler 0.156 μg
Drug: Abediterol 2.5 μg — Dry powder for inhalation
  Arms: Abediterol dry powder inhaler 2.5 μg
Drug: Abediterol 0.05 μg — Pressurised metered-dose inhaler
  Arms: Abediterol pressurised metered-dose inhaler 0.05μg
Drug: Abediterol 0.156 μg — Pressurised metered-dose inhaler
  Arms: Abediterol pressurised metered-dose inhaler 0.156 μg
Drug: Abediterol 2.5 μg — Pressurised metered-dose inhaler
  Arms: Abediterol pressurised metered-dose inhaler 2.5μg
Other: Placebo — Pressurised metered-dose inhaler and dry powder for inhalation.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the pharmacodynamics of single doses of abediterol given by 2 different devices in participants with asthma. Abediterol (AZD0548) is a potential for once daily treatment of asthma and chronic obstructive pulmonary disease (COPD) in fixed dose combination (FDC) with an inhaled corticosteroid (ICS) or a novel anti-inflammatory agent. The aim of the clinical studies is to enable further investigations in participants with asthma and COPD to evaluate and develop abediterol as an effective long acting bronchodilator with an acceptable safety profile compared to other inhaled bronchodilators on the market, for the treatment of asthma and COPD.

DETAILED DESCRIPTION:
This is a randomised, double-blinded, double-dummy, placebo-controlled, multi-centre, six-way William's design, crossover study to assess the pharmacodynamics, pharmacokinetics, and safety of abediterol single dose, given by dry powder inhaler or pressurised metered-dose inhaler, in patients with asthma, on inhaled corticosteroids. During the screening period, all patients will take their own baseline inhaled corticosteroid for 2 weeks. Patients on long-acting β2-agonist/ inhaled corticosteroids will be switched over to the respective inhaled corticosteroid monocomponent. Patients will be provided salbutamol as rescue medication for use throughout the study. Abediterol is an investigational product in early stages of clinical development, therefore individual participants in the clinical studies may not have a clinical benefit, especially in view of alternative therapies (bronchodilators) being available for the treatment of asthma and COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent before any study specific procedures.
2. Men or non-pregnant, non-lactating women 18 to 75 years of age, inclusive.
3. Non-smoker or ex-smoker (quit ≥6months prior to Visit 1) with a total smoking history of ≤10 pack years.
4. Documented clinical diagnosis of asthma for ≥6 months before Visit 1 according to GINA guidelines.
5. On stable dose of ICS or ICS/LABA FDC, for at least 1 month prior to Visit 1, at the doses approved in the country of enrolment.
6. Prebronchodilator FEV1 at Visit 2 ≥40% and ≤85% of predicted (1 repetition of the test is allowed before screen failure).
7. Reversibility to salbutamol (per American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria, 2005 ie, ≥12% and ≥200 mL) at Visit 2 (1 repetition of the test is allowed before screen failure).
8. Demonstrate the ability to use the study inhalation device properly.
9. Able to perform repeated pulmonary function testing for FEV1.
10. Able to read, speak and understand German.
11. Patient must agree to all restrictions during the study.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Participation in another clinical study with an IP during the last 3 months.
3. Known or suspected hypersensitivity to the IP or excipients, including lactose (Note: lactose intolerance is not an exclusion).
4. Systemic steroid use in the 6 weeks before Visit 1.
5. Hospitalization due to asthma in the 6 months prior to Visit 1.
6. Any active pulmonary disease other than asthma.
7. Non-compliance with study procedures in the run in period - as judged by the Investigator.
8. Treatment with biologicals such as monoclonal antibodies or chimeric biomolecules including omalizumab within 6 months or 5 half-lives before Visit 1 (whichever is longer).
9. Treatment with any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to Visit 1.
10. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to Visit 1.
11. Any laboratory abnormality or suspicion of any clinically relevant disease or disorder (on history or examination), including uncontrolled hypertension or uncontrolled diabetes, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study, or any other safety concerns in the opinion of the Investigator.
12. Known chronic hepatitis or HIV infections at the time of enrolment.
13. Any active malignancy or treatment thereof within the 3 years prior to enrolment.
14. Any clinically important abnormalities in rhythm, conduction, or morphology of the screening 12-lead ECG as judged by the Investigator on the screening ECG.
15. Prolonged QT interval using Fridericia's correction 450 msec for males and 470 msec for females on the screening ECG or family history of long QT syndrome.
16. PR (PQ) interval prolongation (> 240 msec), intermittent second or third degree atrialventricular (AV) block or AV dissociation on the screening ECG.
17. Implantable cardiac defibrillator and patients with sustained symptomatic ventricular and/or atrial tachyarrhythmia.
18. Any contraindication against the use of sympathomimetic drugs as judged by the Investigator.
19. Unstable angina pectoris or stable angina pectoris classified higher than Canadian Cardiovascular Society Class II, or a myocardial infarction, or stroke within 6 months before Visit 1.
20. History of hospitalisation within 12 months caused by heart failure or a diagnosis of heart failure higher than New York Heart Association Class II.
21. Suspected poor capability to follow instructions of the study, as judged by the Investigator.
22. History of or current alcohol or drug abuse (including marijuana), as judged by the Investigator.
23. Planned in-patient surgery, major dental procedure or hospitalisation during the study.
24. Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff, contract research organisation staff and/or staff at the study site).
25. Vulnerable persons (eg, persons kept in detention). 26 Daily rescue medication (salbutamol) use of ≥ 12 puffs for ≥ 3 consecutive days during the run-in period.

27. Patient who intends to use any concomitant medication not permitted by this protocol or not to meet the restrictions.

28. Patient on treatment with strong CYP3A4 inhibitors such as ketoconazole or itraconazole or CYP3A4 inducers such as rifampin at Visit 1.

29. Procedures for withdrawal of incorrectly enrolled patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Beier, Dr, Principal Investigator — Biebricher Allee 34, Wiesbaden, Germany, 65187.
Locations (4):
- Germany (4):
  - Research Site, Berlin
  - Research Site, Großhansdorf
  - Research Site, Lübeck
  - Research Site, Wiesbaden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at four sites in Germany.
  The first patient was screened 21 June 2016, the last patient visit was 29 November 2016.
Pre-assignment Details: In total, 42 patients were screened; 30 patients were eligible to participate and were randomised.
Groups:
- Sequence 1: Abediterol dry powder inhaler (DPI) 0.156 μg, followed by Abediterol pressurised metered-dose inhaler (pMDI) 0.05 μg; Placebo; Abediterol pMDI 0.156 μg; Abediterol DPI 2.5 μg; Abediterol pMDI 2.5 μg
- Sequence 2: Abediterol pressurised metered-dose inhaler (pMDI) 0.05 μg, followed by Abediterol pMDI 0.156 μg; Abediterol dry powder inhaler (DPI) 0.156 μg; Abediterol pMDI 2.5 μg; Placebo; Abediterol DPI 2.5 μg
- Sequence 3: Abediterol pressurised metered-dose inhaler (pMDI) 0.156 μg, followed by Abediterol pMDI 2.5 μg; Abediterol pMDI 0.05 μg; Abediterol dry powder inhaler (DPI) 2.5 μg; Abediterol DPI 0.156 μg; Placebo
- Sequence 4: Abediterol dry powder inhaler (DPI) 2.5 μg, followed by Placebo; Abediterol pressurised metered-dose inhaler (pMDI) 2.5 μg; Abediterol DPI 0.156 μg; Abediterol pMDI 0.156 μg; Abediterol pMDI 0.05 μg
- Sequence 5: Abediterol pressurised metered-dose inhaler (pMDI) 2.5 μg, followed by Abediterol dry powder inhaler (DPI) 2.5 μg; Abediterol pMDI 0.156 μg; Placebo; Abediterol pMDI 0.05 μg; Abediterol DPI 0.156 μg
- Sequence 6: Placebo, followed by Abediterol dry powder inhaler (DPI) 0.156 μg; Abediterol DPI 2.5 μg; Abediterol pressurised metered-dose inhaler (pMDI) 0.05 μg; Abediterol pMDI 2.5 μg; Abediterol pMDI 0.156 μg
Period: Treatment Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 4 | 6
Completed | 5 | 5 | 5 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 1 and 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 4 | 6
Completed | 5 | 5 | 5 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 4 | 6
Completed | 5 | 5 | 5 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 2 and 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 4 | 6
Completed | 5 | 5 | 5 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 4 | 6
Completed | 5 | 5 | 5 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 3 and 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 4 | 6
Completed | 5 | 5 | 4 | 5 | 4 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 4 | 5 | 4 | 6
Completed | 5 | 5 | 4 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 4 and 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 4 | 5 | 4 | 6
Completed | 5 | 5 | 4 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 4 | 5 | 4 | 6
Completed | 5 | 5 | 4 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 5 and 6
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 4 | 5 | 4 | 6
Completed | 5 | 5 | 4 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 6
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 4 | 5 | 4 | 6
Completed | 5 | 5 | 4 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all randomised participants who received at least one dose of investigational product
Arm/Group | Overall Study Population
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (10.0)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 10
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1).
Description: Baseline for FEV1 was defined as the mean of the two measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min), prior to the morning investigational product (IP) administration on Day 1 of each treatment period. If both were missing the screening value was used instead.
  Trough is defined as the mean of the FEV1 values obtained at 23 h and 24 h after the morning IP administration. If one of the values was missing, the other one was used as trough.
Time Frame: 45 mins and 15 mins pre-dose, and 23.00-24.00 h post-dose on Day 1
Population: All randomised participants who received investigational product, irrespective of protocol adherence and continued participation in the study
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Liters | 0.225 (0.192) | 0.400 (0.269) | 0.108 (0.212) | 0.170 (0.207) | 0.407 (0.240) | -0.001 (0.244)
Statistical Analysis 1: Comparison: Abediterol Dry Powder Inhaler 0.156 μg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least square mean = 0.2221, 95% CI 2-sided [0.1324 to 0.3118], Standard Error of Mean 0.0453
Statistical Analysis 2: Comparison: Abediterol Dry Powder Inhaler 2.5 μg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean = 0.4042, 95% CI 2-sided [0.3146 to 0.4938], Standard Error of Mean 0.0453
Statistical Analysis 3: Comparison: Abediterol Pressurised Metered-dose Inhaler 0.05μg vs Placebo; Test type: Superiority; p = 0.0207, ANCOVA; Least Square Mean = 0.1056, 95% CI 2-sided [0.0164 to 0.1949], Standard Error of Mean 0.0451
Statistical Analysis 4: Comparison: Abediterol Pressurised Metered-dose Inhaler 0.156 μg vs Placebo; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean = 0.1701, 95% CI 2-sided [0.0810 to 0.2592], Standard Error of Mean 0.0450
Statistical Analysis 5: Comparison: Abediterol Pressurised Metered-dose Inhaler 2.5μg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean = 0.4062, 95% CI 2-sided [0.3170 to 0.4955], Standard Error of Mean 0.0451

2. Secondary Outcome: Percentage of Participants Achieving a ≥ 200 mL and ≥12% Increase From Baseline in Peak FEV1 on Day 1.
Description: The percentage of patients achieving at least 200 mL and 12% increase from baseline in peak FEV1 on Day 1 of each treatment. The peak was the highest value observed during the 6 hour-period immediately after the IP dose in the morning on Day 1.
Time Frame: Predose and 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h and 6 h post-dose on Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Percentage of participants | 72.41 | 82.76 | 56.67 | 73.33 | 90.00 | 24.14

3. Secondary Outcome: Time to Peak FEV1 at Day 1
Description: The peak is the highest forced expiratory volume in one second (FEV1) value observed during the 6 hour-period immediately after the IP dose in the morning on Day 1.
Time Frame: 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h and 6 h post-dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Hours | 3.7 (1.8) | 3.3 (1.8) | 3.0 (1.9) | 3.5 (1.7) | 3.6 (2.0) | 2.9 (2.2)

4. Secondary Outcome: Observed Maximum Concentration of Abediterol (Cmax)
Description: Observed maximum concentration (Cmax) of Abediterol, taken directly from the individual concentration-time curve.
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: The PK analysis set, defined as all randomised subjects who took at least one dose of IP and had at least one evaluable relevant PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 3 | 29 | 0 | 6 | 30 | 0
pg/mL | 0.2299 (117.3) | 1.092 (47.34) |  | 0.2460 (128.7) | 1.211 (82.21) |

5. Secondary Outcome: Time (h) to Maximum Concentration of Abediterol (Tmax).
Description: Time to maximum concentration (Tmax) of Abediterol (h), taken directly from the individual concentration-time curve.
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 3 | 29 | 0 | 6 | 30 | 0
Hours | 0.980 [0.230 to 1.00] | 0.500 [0.230 to 1.00] |  | 0.735 [0.480 to 35.6] | 0.620 [0.070 to 12.0] |

6. Secondary Outcome: Terminal Rate Constant of Abediterol (λz)
Description: Terminal rate constant (λz) of Abediterol, estimated by log-linear least square regression of the terminal part of the concentration-time curve.
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: l/hour
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 0 | 23 | 0 | 0 | 21 | 0
l/hour |  | 0.0526 (0.0228) |  |  | 0.0640 (0.0201) |

7. Secondary Outcome: Terminal Half-life (h) of Abediterol (t½λz)
Description: Terminal half-life (h), estimated as (ln2)/λz (t1/2λz).
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 0 | 23 | 0 | 0 | 21 | 0
Hours |  | 14.99 (4.827) |  |  | 11.85 (3.533) |

8. Secondary Outcome: AUClast of Abediterol
Description: Area under the plasma concentration-curve of Abediterol from time zero to the time of last quantifiable analyte concentration.
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg.h/mL
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 0 | 29 | 0 | 0 | 30 | 0
pg.h/mL |  | 9.092 (53.95) |  |  | 7.674 (132.5) |

9. Secondary Outcome: AUC of Abediterol.
Description: Area under the Abediterol concentration-time curve from time zero extrapolated to infinity (AUC). AUC is estimated by AUClast + Clast/λz where Clast is the last observed quantifiable concentration (AUC).
  PK blood samples were collected 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1 (Note that 24 h and 36 h time-points post-dose correspond to Day 2).
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg.h/mL
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 0 | 23 | 0 | 0 | 21 | 0
pg.h/mL |  | 12.73 (43.26) |  |  | 11.08 (50.01) |

10. Secondary Outcome: Apparent Plasma Clearance for Abediterol (CL/F).
Description: Apparent plasma clearance for parent drug estimated as dose divided by AUC (CL/F).
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 0 | 23 | 0 | 0 | 21 | 0
L/h |  | 196.4 (43.26) |  |  | 225.6 (50.01) |

11. Secondary Outcome: Apparent Volume of Distribution for Abediterol at Terminal Phase (Vz/F).
Description: Apparent volume of distribution for parent drug at terminal phase, estimated by dividing the apparent clearance (CL/F) by λz (Vz/F).
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 0 | 23 | 0 | 0 | 21 | 0
Liters |  | 4008 (37.41) |  |  | 3690 (49.93) |

12. Secondary Outcome: Mean Residence Time (MRT) of Abediterol.
Description: Mean residence time (h), calculated by AUMC/AUC, where AUMC is the area under the first moment-time curve (MRT).
Time Frame: Pre-dose, 5, 15, 30, and 45 minutes, at 1, 2.5, 4, 6, 8, 12, 24 and 36 hours after IP administration on Day 1.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 0 | 23 | 0 | 0 | 21 | 0
Hours |  | 19.73 (35.48) |  |  | 15.59 (29.57) |

13. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event
Description: All treatment emergent adverse events (TEAEs), including serious AEs. An AE is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An AE was considered a TEAE if it was not present prior to the date of the first dose of IP or was present prior to the date of the first dose of IP, but increased in severity after IP administration.
Time Frame: From screening (Day -14) up to follow-up phone call (14 days after last IP administration).
Population: All randomised participants who received at least one dose of investigational product
Measure: Number; unit: Number of participants
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Number of participants | 7 | 10 | 7 | 6 | 7 | 12

14. Secondary Outcome: Number of Participants With Post-baseline Potentially Clinically Significant Abnormalities in Electrocardiogram (ECG) Parameters
Description: Standard 12-lead ECG evaluations were performed prior to IP administration and 1, 4 and 24 h post IP administration at randomisation and after each IP administration. ECGs were recorded after approximately 5 minutes resting in supine position before any blood sampling and spirometry test, preferably always by the same technician for each patient.
  Clinically significant abnormalities were defined as listed in the table below for QT interval, QTcB, QTcF, QRS interval, PR interval and heart rate (HR).
  BL incr. = increase from baseline.
Time Frame: Up to last treatment visit (Day 112)
Population: All randomised participants who received at least one dose of investigational product
Measure: Number; unit: Participants
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Participants
  QT interval >450-<=480msec(Day 1,1h) | 2 | 1 | 2 | 4 | 2 | 3
  QT interval BL incr. >30-<=60msec(Day 1,1h) | 1 | 3 | 0 | 2 | 0 | 4
  QT interval >450-<=480msec(Day 1,4h) | 1 | 1 | 0 | 0 | 2 | 0
  QT interval BL incr. >30-<=60msec(Day 1,4h) | 3 | 3 | 2 | 0 | 1 | 1
  QT interval BL incr. >60msec(Day 1,4h) | 0 | 0 | 0 | 1 | 0 | 0
  QT interval >450-<=480msec(Day 2,24h) | 1 | 0 | 1 | 0 | 1 | 0
  QT interval BL incr. >30-<=60msec(Day 2,24h) | 0 | 1 | 0 | 2 | 1 | 0
  QTcB interval >450-<=480msec(Day 1,1h) | 2 | 1 | 0 | 1 | 1 | 1
  QTcB interval >450-<=480msec(Day 1,4h) | 1 | 2 | 1 | 2 | 1 | 1
  QTcB interval BL incr. >30-<=60msec(Day 1,4h) | 0 | 0 | 0 | 0 | 1 | 0
  QTcB interval >450-<=480msec(Day 2,24h) | 0 | 2 | 1 | 2 | 2 | 2
  QTcB interval BL incr. >30-<=60msec(Day 2,24h) | 0 | 0 | 1 | 0 | 0 | 1
  QTcF interval >450-<=480msec(Day 1,1h) | 0 | 1 | 0 | 2 | 0 | 0
  QTcF interval >450-<=480msec(Day 1,4h) | 0 | 1 | 1 | 1 | 1 | 1
  QTcF interval BL incr. >30-<=60msec(Day 1,4h) | 0 | 1 | 0 | 0 | 0 | 0
  QTcF interval >450-<=480msec(Day 2,24h) | 0 | 1 | 0 | 1 | 0 | 0
  QRS duration >=100 and incr. >=25%(Day 1,4h) | 0 | 0 | 0 | 0 | 1 | 0
  PR interval >=200 and incr. >=25%(Day 1,1h) | 0 | 0 | 0 | 0 | 0 | 1
  PR interval >=200 and incr. >=25%(Day 2,24h) | 0 | 0 | 0 | 0 | 0 | 1
  HR <=50 bpm and decr. >=15%(Day 1,1h) | 1 | 2 | 0 | 4 | 1 | 2
  HR <=50 bpm and decr. >=15%(Day 1,4h) | 1 | 1 | 2 | 2 | 0 | 0
  HR <=50 bpm and decr. >=15%(Day 2,24h) | 0 | 0 | 0 | 1 | 0 | 1

15. Secondary Outcome: Time to Peak FVC at Day 1
Description: The peak is the highest forced vital capacity (FVC) value observed during the 6 hour-period immediately after the IP dose in the morning on Day 1.
Time Frame: 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h and 6 h post-dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Hours | 2.8 (1.8) | 2.3 (1.9) | 2.8 (2.2) | 3.2 (2.3) | 3.4 (2.2) | 1.9 (1.8)

16. Secondary Outcome: Percentage of Participants Achieving a ≥ 200 mL and ≥12% Increase From Baseline in Trough FEV1.
Description: The percentage of patients achieving at least 200 mL and 12% increase from baseline in trough forced expiratory volume in one second (FEV1). Trough was defined as the mean of the FEV1 values obtained at 23 hours and 24 hours after the morning IP administration.
Time Frame: Predose and 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h and 6 h post-dose on Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Percentage of patients | 31.03 | 72.41 | 23.33 | 26.67 | 76.67 | 10.34

17. Secondary Outcome: Change From Baseline in Peak FEV1.
Description: as for outcome 3
Time Frame: Predose and 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h and 6 h post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Liters | 0.4232 (0.0487) | 0.6018 (0.0487) | 0.2930 (0.0483) | 0.4280 (0.0482) | 0.6266 (0.0483) | 0.1880 (0.0486)

18. Secondary Outcome: Change From Baseline in Normalised FEV1 AUC0-24.
Description: Change from baseline in normalised FEV1 area under the concentration-curve of Abediterol from time zero to 24 hours post-dose.
  Baseline for FEV1 was defined as the mean of the 2 measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min before the morning IP administration). If both values were missing, the screening value (pre-bronchodilator FEV1 from Visit 2) was used instead.
Time Frame: 45 mins and 15 mins predose, and 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h, 6 h, 12 h, 16 h, 22 h, and 23.00-24.00 h post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 28
Liters | 0.2767 (0.0468) | 0.4813 (0.0468) | 0.0933 (0.0465) | 0.2091 (0.0464) | 0.4635 (0.0464) | 0.0124 (0.0472)

19. Secondary Outcome: Change From Baseline in Normalised FEV1 AUC0-12.
Description: Change from baseline in normalised FEV1 area under the concentration time curve for Abediterol from time zero to 12 hours post-dose.
  Baseline for FEV1 was defined as the mean of the 2 measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min before the morning IP administration). If both values were missing, the screening value (pre-bronchodilator FEV1 from Visit 2) was used instead.
Time Frame: 45 mins and 15 mins predose, and 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h, 6 h, and 12 h post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 28
Liters | 0.3194 (0.0504) | 0.5135 (0.0504) | 0.1575 (0.0500) | 0.2770 (0.0500) | 0.5104 (0.0500) | 0.0629 (0.0507)

20. Secondary Outcome: Change From Baseline in Normalised FEV1 AUC0-6.
Description: Change from baseline in normalised FEV1 area under the concentration-curve for Abediterol from time zero to 6 hours post-dose.
  Baseline for FEV1 was defined as the mean of the 2 measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min before the morning IP administration). If both values were missing, the screening value (pre-bronchodilator FEV1 from Visit 2) was used instead.
Time Frame: 45 mins and 15 mins predose, and 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h, and 6 h post dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Liters | 0.3198 (0.0485) | 0.5044 (0.0485) | 0.1646 (0.0481) | 0.2987 (0.0480) | 0.5127 (0.0481) | 0.0654 (0.0484)

21. Secondary Outcome: Change From Baseline in Normalised FEV1 AUC12-24.
Description: Change from baseline in normalised FEV1 area under the concentration-curve for Abediterol from time 12 hours post-dose to 24 hours post-dose.
  Baseline for FEV1 was defined as the mean of the 2 measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min before the morning IP administration). If both values were missing, the screening value (pre-bronchodilator FEV1 from Visit 2) was used instead.
Time Frame: 45 mins and 15 mins predose, and 12 h, 16 h, 22 h, and 23.00-24.00 h post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 29 | 30 | 30 | 27
Liters | 0.2339 (0.0479) | 0.4479 (0.0479) | 0.0504 (0.0479) | 0.1421 (0.0474) | 0.4169 (0.0474) | -0.0346 (0.0487)

22. Secondary Outcome: Change From Baseline in Peak FVC.
Description: Baseline for FVC was defined as the mean of the 2 measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min before the morning IP administration). If both values were missing, the screening value (pre-bronchodilator FEV1 from Visit 2) was used instead.
  The peak is the highest forced vital capacity (FVC) value observed during the 6 hour-period immediately after the IP dose in the morning on Day 1.
Time Frame: Predose and 5 mins, 15 mins, 30 mins, 1 h, 2 h, 4 h and 6 h post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Liters | 0.3478 (0.0553) | 0.4932 (0.0552) | 0.2867 (0.0550) | 0.3756 (0.0548) | 0.5059 (0.0549) | 0.2347 (0.0552)

23. Secondary Outcome: Change From Baseline in Trough FVC.
Description: Baseline for FVC was defined as the mean of the two measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min), prior to the morning investigational product (IP)administration on Day 1 of each treatment period. If both were missing the screening value was used instead.
  Trough was defined as the mean of the FEV1 values obtained at 23 h and 24 h after the morning IP administration. If one of the values was missing, the other one was used as trough.
Time Frame: 45 mins and 15 mins pre-dose, and 23.00-24.00 h post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 29
Liters | 0.1702 (0.0523) | 0.3023 (0.0523) | 0.0931 (0.0519) | 0.1218 (0.0517) | 0.3134 (0.0518) | 0.0077 (0.0523)

24. Secondary Outcome: Change From Baseline in Normalised FVC AUC0-24.
Description: Change from baseline in normalised FVC area under the concentration curve for Abediterol from time zero to 24 hours post-dose.
  Baseline for FVC was defined as the mean of the 2 measured values for the corresponding variable (2 measurements 30 min apart, at -45 min and -15 min before the morning IP administration). If both values were missing, the screening value (pre-bronchodilator FVC from Visit 2) was used instead.
Time Frame: as for outcome 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
Number analyzed (Participants) | 29 | 29 | 30 | 30 | 30 | 28
Liters | 0.2057 (0.0513) | 0.3646 (0.0512) | 0.0704 (0.0510) | 0.1445 (0.0508) | 0.3409 (0.0509) | 0.0309 (0.0517)

ADVERSE EVENTS:
Time Frame: From the time of informed consent, throughout the treatment period and including the follow-up period (ie, 2 weeks after last IP dose). Treatment-emergent adverse events were those reported after the first dose of IP up to 30 days after last IP dose.
Description: The safety analysis set consisted of all randomised subjects who received at least one dose of investigational product.
Arm/Group | Abediterol Dry Powder Inhaler 0.156 μg | Abediterol Dry Powder Inhaler 2.5 μg | Abediterol Pressurised Metered-dose Inhaler 0.05μg | Abediterol Pressurised Metered-dose Inhaler 0.156 μg | Abediterol Pressurised Metered-dose Inhaler 2.5μg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/30 | 0/30 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/30 | 0/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 3/29 | 2/29 | 4/30 | 5/30 | 3/30 | 8/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abediterol Dry Powder Inhaler 0.156 μg (N=29) | Abediterol Dry Powder Inhaler 2.5 μg (N=29) | Abediterol Pressurised Metered-dose Inhaler 0.05μg (N=30) | Abediterol Pressurised Metered-dose Inhaler 0.156 μg (N=30) | Abediterol Pressurised Metered-dose Inhaler 2.5μg (N=30) | Placebo (N=29)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 3 (6) | 3 (3) | 3 (4) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Principal Investigator (PI) will be subject to mutual agreement between the PI and the sponsor.